CLINICAL TRIAL: NCT00659152
Title: Morphofunctional Lung Analysis by Positron Emission Tomography in ALI-ARDS Patients
Brief Title: Morphofunctional Lung Analysis by Positron Emission Tomography
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Other Study IDs: 21.02.2008.411
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Acute Lung Injury; Acute Respiratory Distress Syndrome
Keywords: ALI/ARDS
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: ALI/ARDS

SUMMARY:
Patients affected by acute lung injury-acute respiratory distress syndrome (ALI-ARDS) undergo a positron emission tomography (PET) scan in order to analyse lung function.

ELIGIBILITY:
Inclusion Criteria:

* Ali-ards
* Age > 18yrs

Exclusion Criteria:

* COPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALI/ARDS ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Davide Chiumello, Milan, Milano, Italy